CLINICAL TRIAL: NCT04775992
Title: Preemptive Analgesia of Gabapentoids After Major Orthopedic Surgery: Systematic Review and Meta Analysis
Brief Title: Preemptive Analgesia of Gabapentoids in Orthopedic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, SALAH EL-TALLAWY, Professor and Consultant - Anesthesia and Pain Management, King Saud University
Other Study IDs: KSU
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Acute Postoperative Pain
Keywords: acute postoperative pain; Preemptive analgesia; Orthopedic surgery; Preoperative gabapentoids
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preemptive group: patients in this group will receive preoperative gabapentoids
  Interventions: Other: gabapentoids
- control group: patients in this group will not receive gabapentoids
  Interventions: Other: gabapentoids

INTERVENTIONS:
Other: gabapentoids — Preemptive analgesia

SUMMARY:
To address the preemptive analgesic effect of preoperative gabapentoids versus no gabapentoids in orthopedic surgery

DETAILED DESCRIPTION:
Computer search for all studies used preoperative gabapentoids versus no gabapentoids in orthopedic surgery during the last 10 years (from 2011 - 2020)

ELIGIBILITY:
Inclusion Criteria:

* RCT, during last 10 years, involving orthopedic surgery

Exclusion Criteria:

* non randomized trials, unavailable study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all included RCT
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score on rest | every hour for the first 24 hours
  Pain score by VAS on rest
Postoperative pain during movement | every hour for the first 24 hours
  Pain score by VAS during movements

SECONDARY OUTCOMES:
Worst pain score | during the first 24 hours
  Highest pain score
Least pain score | during the first 24 hours
  Lowest pain score
Time spend in severe pain | during the first 24 hours
  how many hours the patients complaint of severe pain
Patient's satisfaction | during the first 24 hours
  Satisfaction by the quality of analgesia

IPD SHARING:
Plan to Share IPD: Undecided